CLINICAL TRIAL: NCT03402880
Title: ALCMI-005: Phase II Study of Pembrolizumab and Epacadostat for Small Cell Lung Cancer After Previous Treatment With Platinum-Based Therapy
Brief Title: ALCMI-005: Pembrolizumab and Epacadostat in Treating Patients With Extensive Stage Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients enrolled
Sponsor: City of Hope Medical Center (Other)
Collaborators: Addario Lung Cancer Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17202; NCI-2017-01756 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2017-11-03; First posted 2018-01-18 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Extensive Stage Small Cell Lung Carcinoma
MeSH Terms: interventions — pembrolizumab; Immunoglobulin G; epacadostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pembrolizumab, epacadostat) (Experimental): Patients receive pembrolizumab IV on day 1 and epacadostat PO BID on days 1-21. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity. Patients benefiting from treatment may continue for an additional 17 courses.
  Interventions: Biological: Pembrolizumab; Drug: Epacadostat; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: 1374853-91-4; Immunoglobulin G4; Anti-(Human Programmed Cell Death 1); Keytruda; Lambrolizumab; MK-3475; SCH 900475; Humanized Mouse Monoclonal (228-L-proline(H10-S>P))gamma 4 Heavy Chain (134-218')-disulfide with Humanized Mouse Monoclonal Kappa Light Chain Dimer (226-226'':229-229'')-bisdisulfide
Drug: Epacadostat — Given PO
  Other Names: INCB024360
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well pembrolizumab and epacadostat work in combination treating patients with extensive stage small cell lung cancer. Monoclonal antibodies, such as pembrolizumab, may assist the immune system in recognizing cancer cells leading to elimination of those cells. Epacadostat may prevent down-regulation of T-cells, which means it can boost the immune system. Giving pembrolizumab and epacadostat together may work better than either drug alone in treating extensive stage small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the objective response rate (ORR) as measured by a modified Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 in subjects with extensive stage small cell lung cancer undergoing treatment with combination pembrolizumab and epacadostat.

SECONDARY OBJECTIVES:

I. To assess the progression free survival (PFS) as measured by a modified RECIST v1.1 in subjects with extensive stage small cell lung cancer undergoing treatment with combination pembrolizumab and epacadostat.

II. To assess the overall survival in subjects with extensive stage small cell lung cancer undergoing treatment with combination pembrolizumab and epacadostat.

III. To assess the >= grade 3 drug related adverse event profile of combination pembrolizumab and epacadostat in subjects with extensive stage small cell lung cancer.

TERTIARY OBJECTIVES:

I. To assess tumor genomics, T-cell, myeloid-derived suppressor cells, and receptors (including PD-L1, IDO1, etc) in relation to response rates.

II. To assess cell free deoxyribonucleic acid (DNA) (cfDNA), cell free ribonucleic acid (RNA) (cfRNA), micro RNA (miRNA), and exosomes as predictors for outcomes to treatment with pembrolizumab and epacadostat in subjects with extensive stage small cell lung cancer and to evaluate plasma for predictive markers for outcomes to therapy.

III. Blood samples will be also be stored for future evaluation.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) on day 1 and epacadostat orally (PO) twice daily (BID) on days 1-21. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity. Patients benefiting from treatment may continue for an additional 17 courses.

After completion of study treatment, patients are followed up at 30 days, then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial
* Subjects with histologically or cytologically confirmed small cell lung cancer and radiographic evidence of extensive stage disease
* Previous treatment with platinum based therapy for small cell lung cancer (eligibility not dependent on stage at time of platinum based therapy)
* Have measurable disease based on RECIST v1.1
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >= 1,500/mcL (performed within 10 days of treatment initiation)
* Platelets >= 100,000/mcL (performed within 10 days of treatment initiation)
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment) (performed within 10 days of treatment initiation)
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) (performed within 10 days of treatment initiation)
* Serum total bilirubin =< 1.2 X ULN OR conjugated bilirubin =< 1.2 x ULN; if an institutional ULN for conjugated bilirubin is not available, then conjugated bilirubin should be < 40% of total bilirubin to be considered eligible (performed within 10 days of treatment initiation)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases (performed within 10 days of treatment initiation)
* Albumin >= 2.5 mg/dL (performed within 10 days of treatment initiation)
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (performed within 10 days of treatment initiation)
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (performed within 10 days of treatment initiation)
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication

  * Note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Male subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

  * Note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy > 10 mg/day prednisone equivalents or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known history of active TB (Bacillus tuberculosis); recommend documentation of inadequate treatment of latent or active TB
* Hypersensitivity to pembrolizumab, epacadostat or any of its excipients
* Corrected QT (QTc) > 480 ms: history or presence of an abnormal electrocardiogram (ECG) that, in the investigators opinion, is clinically meaningful; screening QTc interval > 480 milliseconds is excluded; in the event that a single QTc is > 480 milliseconds, the subject may enroll if the average QTc for the 3 ECGs is < 480 milliseconds; for subjects with an intraventricular conduction delay (QRS interval > 120 milliseconds), the corrected JT (JTc) interval may be used in place of the QTc with sponsor approval; the JTc must be < 340 milliseconds if JTc is used in place of the QTc; subjects with left bundle branch block are excluded; QTc prolongation due to pacemaker may enroll if the JTc is normal
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); exceptions include vitiligo, controlled asthma, type I diabetes, Graves' disease, Hashimoto's disease, or with medical monitor approval; replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Subjects who have had prior radiotherapy within 2 weeks of therapy; subjects must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis; a 1-week wash out is permitted for palliative radiation to non-CNS disease with medical monitor approval
* Has known history of non-infectious pneumonitis that required steroids, evidence of interstitial lung disease or active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Presence of a gastrointestinal condition that may affect drug absorption
* Subjects receiving monoamine oxidase inhibitors (MAOIs) within the 21 days before screening
* Any history of serotonin syndrome after receiving 1 or more serotonergic drugs
* Has a history of other malignancy within 2 years of study entry, with the exception of cured basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive or indolent malignancy, or cancers from which the subject has been disease-free for >= 1 year following treatment with curative intent
* Clinically significant cardiac disease, including unstable angina, acute myocardial infarction within 6 months from day 1 of study drug administration, New York Heart Association class III or IV congestive heart failure, and arrhythmia requiring therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subjects participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-IDO1 agent
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive or hepatitis B virus [HBV] DNA detected) or hepatitis C (e.g., hepatitis C virus [HCV] RNA [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy

  * Note: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate measured by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 | Through study completion, an average of 6 months
  Proportions and associated confidence intervals will be estimated.

SECONDARY OUTCOMES:
Progression free survival | Through study completion, an average of 6 months
  The method of Kaplan-Meier will be used to estimate progression free survival. The Brookmeyer-Crowley method will be used to estimate confidence intervals about median survival times.
Overall survival | Up to 24 months
  The method of Kaplan-Meier will be used to estimate overall survival. The Brookmeyer-Crowley method will be used to estimate confidence intervals about median survival times.
Incidence of grade 3 toxicity | Through study completion, an average of 6 months
  Binary proportions such as toxicity rates can be estimated to within 15% with 95% confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Salgia, MD, Principal Investigator — City of Hope Medical Center; Jacob Sands, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - City of Hope South Pasadena, South Pasadena, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts